CLINICAL TRIAL: NCT04509037
Title: Breast Reductions: Retrospective Evaluation of Suction Assisted Breast Reduction with Peri-Areolar Mastopexy Compared to Longer Incision Pedicle Breast Reduction Techniques
Brief Title: Evaluation of Breast Reduction Techniques
Status: Recruiting | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Herman Houin, MD, Principal Investigator, Henry Ford Health System
Other Study IDs: 7372
Record Dates: First submitted 2020-06-12; First posted 2020-08-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Breast Reductions
Keywords: Breast Reductions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Liposuction Assisted Breast Reduction
- Open Incision Breast Reduction

SUMMARY:
The purpose of this study is to retrospectively evaluate breast reduction techniques in terms of complications, functionality, patient satisfaction, and cosmetic outcomes.

DETAILED DESCRIPTION:
A breast reduction is a common operation with a fairly high complication rate as large incision techniques require undermined skin flaps to be closed under tension. This study is evaluation the open incision breast reduction technique to a liposuction assisted breast reduction. This study will evaluate these two breast reduction techniques in terms of complication rates, functionality, patient satisfaction, and cosmetic outcomes. Participants will be asked to complete the BREAST-Q survey regarding their breast reduction postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a breast reduction between 2013 and 2019
* All patients who underwent a liposuction assisted or layered skin incision pedicled technique breast reduction.

Exclusion Criteria:

* Patients who underwent additional procedures simultaneously at the time of the breast reduction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who underwent a breast reduction between 2013 and 2019.
Sampling Method: Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2012-08-08 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative Complication Rate | Postoperative Period (Average of 1 year following surgery)
  To determine if liposuction assisted breast reduction has a lower postoperative complication rate as opposed to open incision breast reduction
Breast Reduction Success Rate | Postoperative Period (Average of 1 year following surgery)
  To determine if liposuction assisted breast reduction has a higher success rate as opposed to open incision breast reduction based on postoperative outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States